CLINICAL TRIAL: NCT04164095
Title: A Multicenter Randomized Controlled Study of the Effect of Laparoscopic Preservation of the Pylorus and Vagus Nerve on the Postoperative Quality of Life in Patients With Early Gastric Cancer
Brief Title: A Multicenter Randomized Controlled Study of the Effect of Laparoscopic Preservation of the Pylorus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: RenJi Hospital (Other)
Collaborators: The First Affiliated Hospital of Dalian Medical University (Other); Affiliated Hospital of Qinghai University (Other); Zhejiang Cancer Hospital (Other); Second Affiliated Hospital of Suzhou University (Other)
Responsible Party: Principal Investigator, zhaogang, PROFESSOR, RenJi Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LVLM
Record Dates: First submitted 2019-11-12; First posted 2019-11-15 (Actual); Last update posted 2019-12-05 (Actual); Status verified 2019-11

CONDITIONS: Quality of Life

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- lappg (Experimental)
  Interventions: Procedure: lappg
- ladgbi (Active Comparator)
  Interventions: Procedure: lappg

INTERVENTIONS:
Procedure: lappg — Preservation of pylorus and vagus nerve by laparoscopy

SUMMARY:
For the patients with early gastric cancer (T1), preoperative evaluation (gastroscope, ultrasound gastroscope and abdominal enhanced CT) showed that the tumor was located in the body of the stomach, and the margin was enough to retain the pylorus and non lymph node metastasis (N0). Lappg (D1 + lymph node dissection) and traditional laparoscopic distal gastrectomy (BII type anastomosis, D1 + lymph node dissection) were included A control study was conducted to evaluate the influence of two surgical methods on the long-term quality of life of patients after operation

ELIGIBILITY:
Inclusion Criteria:

1. 18 years old < age < 75 years old;
2. primary gastric lesions were diagnosed as gastric adenocarcinoma by biopsy;
3. the preoperative clinical stage was T1N0M0 according to ajcc-7thtnm;
4. it is predicted that R0 can be obtained by pylorogastric gastrectomy and D1 + lymph node dissection;
5. preoperative ECoG physical state score 0 / 1;
6. preoperative ASA score I-III;
7. informed consent of patients.

Exclusion Criteria:

1. pregnant or lactating women; suffering from serious mental illness;
2. the history of upper abdominal surgery (except laparoscopic cholecystectomy);
3. history of gastric surgery (including ESD / EMR for gastric cancer);
4. preoperative imaging examination showed regional enlarged lymph nodes;
5. having other malignant diseases within 5 years;
6. patients with gastric cancer who have received new adjuvant therapy or recommended new adjuvant therapy;
7. there was a history of unstable angina or myocardial infarction within 6 months;
8. have a history of cerebral infarction or cerebral hemorrhage within 6 months;
9. there was a history of continuous systemic corticosteroid therapy within 1 month;
10. simultaneous surgical treatment of other diseases is needed;
11. gastric cancer with complications (hemorrhage, perforation, obstruction) requires emergency surgery;
12. FEV1 of pulmonary function examination was less than 50% of the predicted value.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2020-01-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
EORTC-QLQ-C30 | 5 years
  score: 0-100. more global and functional scales is better. less symptom scales is better

IPD SHARING:
Plan to Share IPD: Undecided